CLINICAL TRIAL: NCT05780047
Title: Personalized Mobile Intervention to Reduce Exposure to Endocrine Disrupting Chemicals (EDCs) in Women of Child-Bearing Age and Their Partners
Brief Title: Personalized Mobile Intervention to Reduce Exposure to Endocrine Disrupting Chemicals in Adults of Child-Bearing Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Million Marker Wellness, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R43ES034312-01 (NIH)
Record Dates: First submitted 2023-02-27; First posted 2023-03-22 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Endocrine Disrupting Chemicals; Environmental Exposure; Health Literacy; Bisphenol A; Phthalate Exposure; Survey
Keywords: parabens; exposure; environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile EDC reduction program (Experimental): Million Marker's (MM) first-of-its-kind mobile endocrine disrupting chemical (EDC) reduction program will be tested and validated in a prospective longitudinal cohort intervention trial. 50 women in reproductive age and their partners will be recruited from the Healthy Nevada Project, an existing state-wide health monitoring effort. Using MM's services, participants' urine samples will be collected two times (at pre- and post-intervention) to measure changes in EDC levels. Changes in participants' environmental health literacy, attitudes, knowledge, and behaviors will be assessed after using MM's products and services. Validated surveys on environmental health literacy and readiness to change and analyses of participants' lifestyle behaviors and product use will be conducted at baseline (first test) and upon completion of the second test. The investigators will evaluate the MM app and platform usability to improve the user experience, using the System Usability Score (SUS) survey.
  Interventions: Diagnostic Test: Mail-in Urine Test for EDCs

INTERVENTIONS:
Diagnostic Test: Mail-in Urine Test for EDCs — Million Marker provides a mail-in urine test for Bisphenol A (BPA) and phthalates. Users take a comprehensive exposure survey (via the MM app), send back their samples, view their personalized reports with tailored product recommendations, make changes to reduce their exposures, and retest to monitor their progress. Participants will also fill out surveys to assess changes in their environmental health literacy, readiness to change, and analyses of lifestyle behaviors and product use.
  Other Names: Million Marker Detect and Detox test kit

SUMMARY:
The goal of this intervention study is to determine to what extent the Million Marker (MM) program reduces users' endocrine disruption chemical (EDC) exposure levels and changes their environmental health awareness and behaviors. The main questions it aims to answer are:

* Can the investigators see a reduction in EDC levels in participants' urine samples after using the MM Detect and Detox kit?
* Can the investigators see a change in participants' environmental health literacy, knowledge, and behaviors after using MM's products and services?
* How can Million Marker improve their app and platform to improve the user experience? Participants will collect their urine pre- and post-intervention, and will take a comprehensive exposure survey (via the MM app) before sending back their samples. This exposure survey will ask about participant's product use, diet, and lifestyle behaviors. Participants will also fill out surveys pre- and post-intervention assessing their perception of environmental health, as well as usability of the platform.

DETAILED DESCRIPTION:
Exposures to endocrine disrupting chemicals (EDCs) have been linked to chronic diseases and conditions including breast cancer, metabolic syndrome, diabetes, and infertility. Timing of exposure, especially during pregnancy, may have a lifelong impact on the fetus, including neurodevelopmental problems and asthma. However, there have been no tools to allow those in the preconception, conception, and pregnancy stages to assess EDC exposures to ensure a healthy pregnancy and normal child development. Million Marker (MM) was born to fill this need. MM is a precision health company, built by a team of multidisciplinary scientists who are trained in environmental epidemiology, toxicology, analytical chemistry, biostatistics, data engineering, and business. MM's missions are to crowdsource and scale the biomonitoring of environmental chemicals and provide actionable results to consumers in a timely manner in order to empower individuals to proactively assess, track, and reduce their harmful environmental exposures. Starting with a few biomarkers of common EDCs, MM's ultimate vision is to discover all possible ("a million") biomarkers of harmful exposures to inform and improve individual health outcomes and advance precision medicine. Less than a year after it was founded, Million Marker developed and sold the first product-a mail-in urine test for BPA and phthalates-and successfully helped users reduce exposures through personalized intervention plans. Customers are able to order a test kit online, receive the test kit via mail, take a comprehensive exposure survey (via the Million Marker app), send back samples via mail, view personalized reports with tailored product recommendations through a secure online portal, make lifestyle changes to reduce exposures, and retest to monitor progress. MM's initial target audience are individuals of reproductive age, due to the vulnerability pregnancy and preconception to EDC exposures. However, it is unclear to what extent the MM platform educates, motivates, and ultimately reduces EDC exposure in individuals in this age range. Therefore, the aims of the current proposal are to 1) test and validate a this first-of-its-kind mobile EDC reduction program in a prospective longitudinal cohort intervention trial; 2) assess changes in participants' environmental health literacy, attitudes, knowledge, and behaviors after using MM's products and services; and 3) evaluate the MM app and platform usability to improve the user experience. Validating this population with MM's program is a step towards these types of future studies. At the conclusion of the project, MM will be well-positioned to begin Phase II and will scale the EDCs testing and personalized intervention plan to fertility clinics and the general public.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-40 years
* in good health, not pregnant, free from diabetes or known kidney disease or cancer (these conditions may interfere with EDC metabolism)
* able to understand written and spoken English
* already consented for re-contact with the Healthy Nevada Project
* owning a smartphone
* willing to complete all study assessments

Exclusion Criteria:

* only one woman and her partner per household will be enrolled

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 434 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hua, PhD, Principal Investigator — Million Marker Wellness, Inc.
Locations (1):
- Million Marker Wellness Inc., Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Million Marker will disseminate research results and findings to the scientific community through presentations at scientific meetings and conferences and publications in academic journals, as well as through the mass media and online postings. The Principal Investigator of this study will make data and associated documentation/metadata available to external researchers under a data-sharing agreement in which a specific commitment is made to use the data for research purposes only, to not provide the data to a third party or distribute it in any form, and to properly acknowledge the source of funding for the collection of the data and the researchers involved in this study.
Time Frame: Starting 6 months after publication
Access Criteria: Researchers must submit an acceptable research plan (goals of the proposed research, the specific hypotheses to be examined, justification for research and methods), be affiliated with a recognized research institution, have demonstrated expertise in the area of the proposed research project, and receive independent approval from their governing institutional review board. Data will be available for use only to answer the specific question(s) indicated in the research plan. The researchers must provide a list of variable names and an outline of how research findings will be disseminated; and will be asked to sign a data-sharing agreement that commits to: 1) not attempt to identify any individual participant, 2) secure the data using appropriate software technology, 3) and destroy or return all data once analyses are complete. All final datasets will be de-identified. Final authorship on manuscripts will require review and approval by the Principal Investigators of this study.

REFERENCES:
- [Background] Bowes DA, Halden RU. Breast Cancer and Dietary Intake of Endocrine Disruptors: a Review of Recent Literature. Curr. Pathobiol. Rep. 2019; 7:41-46.
- [Background] Hiatt RA, Brody JG. Environmental Determinants of Breast Cancer. Annu Rev Public Health. 2018 Apr 1;39:113-133. doi: 10.1146/annurev-publhealth-040617-014101. Epub 2018 Jan 12. PMID 29328875
- [Background] Heindel JJ, Blumberg B, Cave M, Machtinger R, Mantovani A, Mendez MA, Nadal A, Palanza P, Panzica G, Sargis R, Vandenberg LN, Vom Saal F. Metabolism disrupting chemicals and metabolic disorders. Reprod Toxicol. 2017 Mar;68:3-33. doi: 10.1016/j.reprotox.2016.10.001. Epub 2016 Oct 17. PMID 27760374
- [Background] Hwang S, Lim JE, Choi Y, Jee SH. Bisphenol A exposure and type 2 diabetes mellitus risk: a meta-analysis. BMC Endocr Disord. 2018 Nov 6;18(1):81. doi: 10.1186/s12902-018-0310-y. PMID 30400886
- [Background] Ghayda RA, Williams PL, Chavarro JE, Ford JB, Souter I, Calafat AM, Hauser R, Minguez-Alarcon L. Urinary bisphenol S concentrations: Potential predictors of and associations with semen quality parameters among men attending a fertility center. Environ Int. 2019 Oct;131:105050. doi: 10.1016/j.envint.2019.105050. Epub 2019 Jul 31. PMID 31376593
- [Background] Machtinger R, Gaskins AJ, Racowsky C, Mansur A, Adir M, Baccarelli AA, Calafat AM, Hauser R. Urinary concentrations of biomarkers of phthalates and phthalate alternatives and IVF outcomes. Environ Int. 2018 Feb;111:23-31. doi: 10.1016/j.envint.2017.11.011. Epub 2017 Nov 20. PMID 29161633
- [Background] Braun JM. Early-life exposure to EDCs: role in childhood obesity and neurodevelopment. Nat Rev Endocrinol. 2017 Mar;13(3):161-173. doi: 10.1038/nrendo.2016.186. Epub 2016 Nov 18. PMID 27857130
- [Background] Mustieles V, Zhang Y, Yland J, Braun JM, Williams PL, Wylie BJ, Attaman JA, Ford JB, Azevedo A, Calafat AM, Hauser R, Messerlian C. Maternal and paternal preconception exposure to phenols and preterm birth. Environ Int. 2020 Apr;137:105523. doi: 10.1016/j.envint.2020.105523. Epub 2020 Feb 29. PMID 32120140
- [Background] Woods MM, Lanphear BP, Braun JM, McCandless LC. Gestational exposure to endocrine disrupting chemicals in relation to infant birth weight: a Bayesian analysis of the HOME Study. Environ Health. 2017 Oct 27;16(1):115. doi: 10.1186/s12940-017-0332-3. PMID 29078782
- [Background] Veiga-Lopez A, Kannan K, Liao C, Ye W, Domino SE, Padmanabhan V. Gender-Specific Effects on Gestational Length and Birth Weight by Early Pregnancy BPA Exposure. J Clin Endocrinol Metab. 2015 Nov;100(11):E1394-403. doi: 10.1210/jc.2015-1724. Epub 2015 Sep 25. PMID 26406292
- [Background] Raghavan R, Romano ME, Karagas MR, Penna FJ. Pharmacologic and Environmental Endocrine Disruptors in the Pathogenesis of Hypospadias: a Review. Curr Environ Health Rep. 2018 Dec;5(4):499-511. doi: 10.1007/s40572-018-0214-z. PMID 30578470
- [Background] Gascon M, Casas M, Morales E, Valvi D, Ballesteros-Gomez A, Luque N, Rubio S, Monfort N, Ventura R, Martinez D, Sunyer J, Vrijheid M. Prenatal exposure to bisphenol A and phthalates and childhood respiratory tract infections and allergy. J Allergy Clin Immunol. 2015 Feb;135(2):370-8. doi: 10.1016/j.jaci.2014.09.030. Epub 2014 Oct 30. PMID 25445825
- [Background] Paciencia I, Cavaleiro Rufo J, Silva D, Martins C, Mendes F, Farraia M, Delgado L, de Oliveira Fernandes E, Padrao P, Moreira P, Severo M, Barros H, Moreira A. Exposure to indoor endocrine-disrupting chemicals and childhood asthma and obesity. Allergy. 2019 Jul;74(7):1277-1291. doi: 10.1111/all.13740. Epub 2019 Mar 5. PMID 30740706
- [Background] Kalkbrenner AE, Schmidt RJ, Penlesky AC. Environmental chemical exposures and autism spectrum disorders: a review of the epidemiological evidence. Curr Probl Pediatr Adolesc Health Care. 2014 Nov;44(10):277-318. doi: 10.1016/j.cppeds.2014.06.001. Epub 2014 Sep 5. PMID 25199954
- [Background] Oulhote Y, Lanphear B, Braun JM, Webster GM, Arbuckle TE, Etzel T, Forget-Dubois N, Seguin JR, Bouchard MF, MacFarlane A, Ouellet E, Fraser W, Muckle G. Gestational Exposures to Phthalates and Folic Acid, and Autistic Traits in Canadian Children. Environ Health Perspect. 2020 Feb;128(2):27004. doi: 10.1289/EHP5621. Epub 2020 Feb 19. PMID 32073305
- [Background] Gutierrez-Torres DS, Barraza-Villarreal A, Hernandez-Cadena L, Escamilla-Nunez C, Romieu I. Prenatal Exposure to Endocrine Disruptors and Cardiometabolic Risk in Preschoolers: A Systematic Review Based on Cohort Studies. Ann Glob Health. 2018 Jul 27;84(2):239-249. doi: 10.29024/aogh.911. PMID 30873814
- [Background] American College of Obstetricians and Gynecologists' Committee on Obstetric Practice. Reducing Prenatal Exposure to Toxic Environmental Agents: ACOG Committee Opinion, Number 832. Obstet Gynecol. 2021 Jul 1;138(1):e40-e54. doi: 10.1097/AOG.0000000000004449. PMID 34259492
- [Background] NCHS. National Health and Nutrition Examination Survey Overview. 2020. https://www.cdc.gov/nchs/data/nhanes/nhanes_13_14/NHANES_Overview_Brochure.pdf
- [Background] Birnbaum LS, Jung P. From endocrine disruptors to nanomaterials: advancing our understanding of environmental health to protect public health. Health Aff (Millwood). 2011 May;30(5):814-22. doi: 10.1377/hlthaff.2010.1225. PMID 21555467
- [Background] Walker DI, Valvi D, Rothman N, Lan Q, Miller GW, Jones DP. The metabolome: A key measure for exposome research in epidemiology. Curr Epidemiol Rep. 2019;6:93-103. Epub 2019 Apr 26. PMID 31828002
- [Background] Google. Google Trends 'Chemical Free' 2004-present. 2020. https://trends.google.com/trends/explore?date=all&geo=US&q=%2Fm%2F09gd7dm
- [Background] Rock Health. Healthcare consumers in a digital transition. Results from our third national consumer survey (2017 data) on digital health adoption and sentiments. 2020. https://rockhealth.com/reports/healthcare-consumers-in-a-digital-transition/
- [Background] Rappaport SM, Smith MT. Epidemiology. Environment and disease risks. Science. 2010 Oct 22;330(6003):460-1. doi: 10.1126/science.1192603. PMID 20966241
- [Background] Calkins K, Devaskar SU. Fetal origins of adult disease. Curr Probl Pediatr Adolesc Health Care. 2011 Jul;41(6):158-76. doi: 10.1016/j.cppeds.2011.01.001. PMID 21684471
- [Background] Wild CP. Complementing the genome with an "exposome": the outstanding challenge of environmental exposure measurement in molecular epidemiology. Cancer Epidemiol Biomarkers Prev. 2005 Aug;14(8):1847-50. doi: 10.1158/1055-9965.EPI-05-0456. No abstract available. PMID 16103423
- [Background] Wild CP. The exposome: from concept to utility. Int J Epidemiol. 2012 Feb;41(1):24-32. doi: 10.1093/ije/dyr236. Epub 2012 Jan 31. No abstract available. PMID 22296988
- [Background] CDC. NHANES: National Health and Nutrition Examination Survey. 2020. https://www.cdc.gov/nchs/nhanes/index.htm
- [Background] CDC. State Biomonitoring Programs. National Biomonitoring Program. 2019. https://www.cdc.gov/biomonitoring/state_grants.html
- [Background] CDC. Updated Tables, January 2019. National Report on Human Exposure to Environmental Chemicals. 2019. https://www.cdc.gov/exposurereport/index.html
- [Background] CDC. National Center for Health Statistics National Health and Nutrition Examination Survey Overview. https://www.cdc.gov/nchs/data/nhanes/nhanes_13_14/NHANES_Overview_Brochure.pdf.
- [Background] Dennis KK, Marder E, Balshaw DM, Cui Y, Lynes MA, Patti GJ, Rappaport SM, Shaughnessy DT, Vrijheid M, Barr DB. Biomonitoring in the Era of the Exposome. Environ Health Perspect. 2017 Apr;125(4):502-510. doi: 10.1289/EHP474. Epub 2016 Jul 6. PMID 27385067
- [Background] Rochester JR. Bisphenol A and human health: a review of the literature. Reprod Toxicol. 2013 Dec;42:132-55. doi: 10.1016/j.reprotox.2013.08.008. Epub 2013 Aug 30. PMID 23994667
- [Background] Paulose T, Speroni L, Sonnenschein C, Soto AM. Estrogens in the wrong place at the wrong time: Fetal BPA exposure and mammary cancer. Reprod Toxicol. 2015 Jul;54:58-65. doi: 10.1016/j.reprotox.2014.09.012. Epub 2014 Sep 30. PMID 25277313
- [Background] Street ME, Angelini S, Bernasconi S, Burgio E, Cassio A, Catellani C, Cirillo F, Deodati A, Fabbrizi E, Fanos V, Gargano G, Grossi E, Iughetti L, Lazzeroni P, Mantovani A, Migliore L, Palanza P, Panzica G, Papini AM, Parmigiani S, Predieri B, Sartori C, Tridenti G, Amarri S. Current Knowledge on Endocrine Disrupting Chemicals (EDCs) from Animal Biology to Humans, from Pregnancy to Adulthood: Highlights from a National Italian Meeting. Int J Mol Sci. 2018 Jun 2;19(6):1647. doi: 10.3390/ijms19061647. PMID 29865233
- [Background] Trasande L, Zoeller RT, Hass U, Kortenkamp A, Grandjean P, Myers JP, DiGangi J, Hunt PM, Rudel R, Sathyanarayana S, Bellanger M, Hauser R, Legler J, Skakkebaek NE, Heindel JJ. Burden of disease and costs of exposure to endocrine disrupting chemicals in the European Union: an updated analysis. Andrology. 2016 Jul;4(4):565-72. doi: 10.1111/andr.12178. Epub 2016 Mar 22. PMID 27003928
- [Background] CDC. Bisphenol A (BPA) Factsheet. National Biomonitoring Program. 2017. https://www.cdc.gov/biomonitoring/BisphenolA_FactSheet.html
- [Background] Harley KG, Kogut K, Madrigal DS, Cardenas M, Vera IA, Meza-Alfaro G, She J, Gavin Q, Zahedi R, Bradman A, Eskenazi B, Parra KL. Reducing Phthalate, Paraben, and Phenol Exposure from Personal Care Products in Adolescent Girls: Findings from the HERMOSA Intervention Study. Environ Health Perspect. 2016 Oct;124(10):1600-1607. doi: 10.1289/ehp.1510514. Epub 2016 Mar 7. PMID 26947464
- [Background] Kelley AS, Banker M, Goodrich JM, Dolinoy DC, Burant C, Domino SE, Smith YR, Song PXK, Padmanabhan V. Early pregnancy exposure to endocrine disrupting chemical mixtures are associated with inflammatory changes in maternal and neonatal circulation. Sci Rep. 2019 Apr 1;9(1):5422. doi: 10.1038/s41598-019-41134-z. PMID 30931951
- [Background] Attina TM, Hauser R, Sathyanarayana S, Hunt PA, Bourguignon JP, Myers JP, DiGangi J, Zoeller RT, Trasande L. Exposure to endocrine-disrupting chemicals in the USA: a population-based disease burden and cost analysis. Lancet Diabetes Endocrinol. 2016 Dec;4(12):996-1003. doi: 10.1016/S2213-8587(16)30275-3. Epub 2016 Oct 17. PMID 27765541
- [Background] WHO. Human Biomonitoring: Facts and Figures. 2015. http://www.euro.who.int/__data/assets/pdf_file/0020/276311/Human-biomonitoring-facts-figures-en.pdf
- [Background] Bocato MZ, Bianchi Ximenez JP, Hoffmann C, Barbosa F. An overview of the current progress, challenges, and prospects of human biomonitoring and exposome studies. J Toxicol Environ Health B Crit Rev. 2019;22(5-6):131-156. doi: 10.1080/10937404.2019.1661588. Epub 2019 Sep 5. PMID 31543064
- [Background] Pew Research Center. Mobile Fact Sheet. Internet & Technology. 2019. https://www.pewresearch.org/internet/fact-sheet/mobile/
- [Background] Apple Inc. App Store. 2020. https://www.apple.com/ios/app-store/
- [Background] Google. Google Play Store. 2020. https://play.google.com/store?hl=en_US
- [Background] Han M, Lee E. Effectiveness of Mobile Health Application Use to Improve Health Behavior Changes: A Systematic Review of Randomized Controlled Trials. Healthc Inform Res. 2018 Jul;24(3):207-226. doi: 10.4258/hir.2018.24.3.207. Epub 2018 Jul 31. PMID 30109154
- [Background] Sawesi S, Rashrash M, Phalakornkule K, Carpenter JS, Jones JF. The Impact of Information Technology on Patient Engagement and Health Behavior Change: A Systematic Review of the Literature. JMIR Med Inform. 2016 Jan 21;4(1):e1. doi: 10.2196/medinform.4514. PMID 26795082
- [Background] Michie S, Yardley L, West R, Patrick K, Greaves F. Developing and Evaluating Digital Interventions to Promote Behavior Change in Health and Health Care: Recommendations Resulting From an International Workshop. J Med Internet Res. 2017 Jun 29;19(6):e232. doi: 10.2196/jmir.7126. PMID 28663162
- [Background] Partridge SR, Redfern J. Strategies to Engage Adolescents in Digital Health Interventions for Obesity Prevention and Management. Healthcare (Basel). 2018 Jun 21;6(3):70. doi: 10.3390/healthcare6030070. PMID 29933550
- [Background] Milne-Ives M, Lam C, Van Velthoven MH, Meinert E. Mobile Apps for Health Behavior Change: Protocol for a Systematic Review. JMIR Res Protoc. 2020 Jan 30;9(1):e16931. doi: 10.2196/16931. PMID 32012109
- [Background] Oikonomidi T, Vivot A, Tran VT, Riveros C, Robin E, Ravaud P. A Methodologic Systematic Review of Mobile Health Behavior Change Randomized Trials. Am J Prev Med. 2019 Dec;57(6):836-843. doi: 10.1016/j.amepre.2019.07.008. PMID 31753266
- [Background] Carwile JL, Ye X, Zhou X, Calafat AM, Michels KB. Canned soup consumption and urinary bisphenol A: a randomized crossover trial. JAMA. 2011 Nov 23;306(20):2218-20. doi: 10.1001/jama.2011.1721. No abstract available. PMID 22110104
- [Background] Rudel RA, Gray JM, Engel CL, Rawsthorne TW, Dodson RE, Ackerman JM, Rizzo J, Nudelman JL, Brody JG. Food packaging and bisphenol A and bis(2-ethyhexyl) phthalate exposure: findings from a dietary intervention. Environ Health Perspect. 2011 Jul;119(7):914-20. doi: 10.1289/ehp.1003170. Epub 2011 Mar 30. PMID 21450549
- [Background] Peng CY, Tsai EM, Kao TH, Lai TC, Liang SS, Chiu CC, Wang TN. Canned food intake and urinary bisphenol a concentrations: a randomized crossover intervention study. Environ Sci Pollut Res Int. 2019 Sep;26(27):27999-28009. doi: 10.1007/s11356-019-05534-y. Epub 2019 Jul 27. PMID 31352597
- [Background] Ji K, Lim Kho Y, Park Y, Choi K. Influence of a five-day vegetarian diet on urinary levels of antibiotics and phthalate metabolites: a pilot study with "Temple Stay" participants. Environ Res. 2010 May;110(4):375-82. doi: 10.1016/j.envres.2010.02.008. Epub 2010 Mar 12. PMID 20227070
- [Background] Chen CY, Chou YY, Lin SJ, Lee CC. Developing an intervention strategy to reduce phthalate exposure in Taiwanese girls. Sci Total Environ. 2015 Jun 1;517:125-31. doi: 10.1016/j.scitotenv.2015.02.021. Epub 2015 Feb 25. PMID 25725197
- [Background] Sathyanarayana S, Alcedo G, Saelens BE, Zhou C, Dills RL, Yu J, Lanphear B. Unexpected results in a randomized dietary trial to reduce phthalate and bisphenol A exposures. J Expo Sci Environ Epidemiol. 2013 Jul;23(4):378-84. doi: 10.1038/jes.2013.9. Epub 2013 Feb 27. PMID 23443238
- [Background] Guo W, Huen K, Park JS, Petreas M, Crispo Smith S, Block G, Holland N. Vitamin C intervention may lower the levels of persistent organic pollutants in blood of healthy women - A pilot study. Food Chem Toxicol. 2016 Jun;92:197-204. doi: 10.1016/j.fct.2016.04.006. Epub 2016 Apr 23. PMID 27090108
- [Background] Correia-Sa L, Kasper-Sonnenberg M, Palmke C, Schutze A, Norberto S, Calhau C, Domingues VF, Koch HM. Obesity or diet? Levels and determinants of phthalate body burden - A case study on Portuguese children. Int J Hyg Environ Health. 2018 Apr;221(3):519-530. doi: 10.1016/j.ijheh.2018.02.001. Epub 2018 Feb 6. PMID 29454883
- [Background] Galloway TS, Baglin N, Lee BP, Kocur AL, Shepherd MH, Steele AM; BPA Schools Study Consortium; Harries LW. An engaged research study to assess the effect of a 'real-world' dietary intervention on urinary bisphenol A (BPA) levels in teenagers. BMJ Open. 2018 Feb 3;8(2):e018742. doi: 10.1136/bmjopen-2017-018742. PMID 29431133
- [Background] Hagobian T, Smouse A, Streeter M, Wurst C, Schaffner A, Phelan S. Randomized Intervention Trial to Decrease Bisphenol A Urine Concentrations in Women: Pilot Study. J Womens Health (Larchmt). 2017 Feb;26(2):128-132. doi: 10.1089/jwh.2016.5746. Epub 2016 Oct 11. PMID 27726525
- [Background] Hyland C, Bradman A, Gerona R, Patton S, Zakharevich I, Gunier RB, Klein K. Organic diet intervention significantly reduces urinary pesticide levels in U.S. children and adults. Environ Res. 2019 Apr;171:568-575. doi: 10.1016/j.envres.2019.01.024. Epub 2019 Feb 12. PMID 30765100
- [Background] Ackerman JM, Dodson RE, Engel CL, Gray JM, Rudel RA. Temporal variability of urinary di(2-ethylhexyl) phthalate metabolites during a dietary intervention study. J Expo Sci Environ Epidemiol. 2014 Nov;24(6):595-601. doi: 10.1038/jes.2013.93. Epub 2014 Jan 22. PMID 24448002
- [Background] Grzymski, J. J. et al. The Healthy Nevada Project: rapid recruitment for population health study. 2018. http://biorxiv.org/lookup/doi/10.1101/250274. doi:10.1101/250274.
- [Background] Healthy Nevada Project. About Us. https://healthynv.org/about/.
- [Background] CDC. Fourth National Report on Human Exposure to Environmental Chemicals, Updated Tables, January 2019, Volume 2. 2019. https://www.cdc.gov/exposurereport/pdf/FourthReport_UpdatedTables_Volume2_Jan2019-508.pdf
- [Background] Lehmler HJ, Liu B, Gadogbe M, Bao W. Exposure to Bisphenol A, Bisphenol F, and Bisphenol S in U.S. Adults and Children: The National Health and Nutrition Examination Survey 2013-2014. ACS Omega. 2018 Jun 30;3(6):6523-6532. doi: 10.1021/acsomega.8b00824. Epub 2018 Jun 18. PMID 29978145
- [Background] Meeker JD, Ferguson KK. Urinary phthalate metabolites are associated with decreased serum testosterone in men, women, and children from NHANES 2011-2012. J Clin Endocrinol Metab. 2014 Nov;99(11):4346-52. doi: 10.1210/jc.2014-2555. Epub 2014 Aug 14. PMID 25121464
- [Background] Calafat AM, Ye X, Wong LY, Bishop AM, Needham LL. Urinary concentrations of four parabens in the U.S. population: NHANES 2005-2006. Environ Health Perspect. 2010 May;118(5):679-85. doi: 10.1289/ehp.0901560. Epub 2010 Jan 4. PMID 20056562
- [Background] Calafat AM, Wong LY, Ye X, Reidy JA, Needham LL. Concentrations of the sunscreen agent benzophenone-3 in residents of the United States: National Health and Nutrition Examination Survey 2003--2004. Environ Health Perspect. 2008 Jul;116(7):893-7. doi: 10.1289/ehp.11269. PMID 18629311
- [Background] Lichtveld MY, Covert HH, Sherman M, Shankar A, Wickliffe JK, Alcala CS. Advancing Environmental Health Literacy: Validated Scales of General Environmental Health and Environmental Media-Specific Knowledge, Attitudes and Behaviors. Int J Environ Res Public Health. 2019 Oct 28;16(21):4157. doi: 10.3390/ijerph16214157. PMID 31661913
- [Background] American Council on Exercise. Readiness to Change Questionnaire. 2014.
- [Background] van der Vaart R, Drossaert C. Development of the Digital Health Literacy Instrument: Measuring a Broad Spectrum of Health 1.0 and Health 2.0 Skills. J Med Internet Res. 2017 Jan 24;19(1):e27. doi: 10.2196/jmir.6709. PMID 28119275
- [Background] U.S. Department of Health and Human Services. System Usability Scale (SUS). 2020. https://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2021 and July 2022, recruitment emails describing the study and asking for participation were sent to Healthy Nevada Project participants.
Groups:
- Mobile EDC Reduction Program: Million Marker's (MM) mobile endocrine disrupting chemical (EDC) reduction program will be tested and validated in a prospective longitudinal cohort intervention trial. 50 women in reproductive age and their partners will be recruited from the Healthy Nevada Project, an existing state-wide health monitoring effort. Using MM's services, participants' urine samples will be collected two times (at pre- and post-intervention) to measure changes in EDC levels. Changes in participants' environmental health literacy, attitudes, knowledge, and behaviors will be assessed after using MM's products and services. Validated surveys on environmental health literacy and readiness to change and analyses of participants' lifestyle behaviors and product use will be conducted at baseline and upon completion of the second test. The investigators will evaluate the MM app and platform usability to improve the user experience, using the System Usability Score (SUS) survey.
  Mail-in Urine Test for EDCs: Million Marker provides a mail-in urine test for Bisphenol A (BPA) and phthalates. Users take a comprehensive exposure survey (via the MM app), send back their samples, view their personalized reports with tailored product recommendations, make changes to reduce their exposures, and retest to monitor their progress. Participants will also fill out surveys to assess changes in their environmental health literacy, readiness to change, and analyses of lifestyle behaviors and product use.
Period: Overall Study
Arm/Group | Mobile EDC Reduction Program
Started | 434
Completed | 50
Not Completed | 384
Not completed — Did not submit baseline urine test kit | 226
Not completed — Lost to Follow-up | 34
Not completed — Did not submit second urine test kit | 124

BASELINE CHARACTERISTICS:
Arm/Group | Mobile EDC Reduction Program
Number analyzed (Participants) | 434
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 434
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 30.7 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants did not enter their age in the survey (missing data).
  Participants
    number analyzed (Participants) | 432
    Female | 328
    Male | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12
  Black | 2
  Hispanic or Latino | 44
  Native American | 3
  Pacific Islander | 7
  White | 344
  Other | 22
Region of Enrollment [Number; unit: participants] — Participants were recruited through the Healthy Nevada Project which serves Northern Nevada, US
  participants
    United States | 434
Baseline metabolite concentrations [Mean (Standard Deviation); unit: ng/ml] — Population: Only 208 participants returned baseline urine test kits and 17 kits had errors in the lab analyses, resulting in 191 participants with baseline metabolite values.
  ng/ml
    methyl paraben: number analyzed (Participants) | 191
    methyl paraben | 69.48 (215.69)
    propyl paraben: number analyzed (Participants) | 191
    propyl paraben | 22.86 (87.07)
    monobutyl phthalate: number analyzed (Participants) | 191
    monobutyl phthalate | 71.52 (105.73)
    monoethyl phthalate: number analyzed (Participants) | 191
    monoethyl phthalate | 151.60 (442.17)
    mono-(2-ethyl-5-carboxypentyl) phthalate: number analyzed (Participants) | 191
    mono-(2-ethyl-5-carboxypentyl) phthalate | 5.32 (17.88)
Environmental Health Literacy [Mean (Standard Deviation); unit: Scores on a Likert scale] — Validated survey on environmental health literacy will be conducted at baseline and upon completion of the second test. The surveys will be compared for changes. The EHL survey was adapted from the "General Environmental Health Scale" with three subscales: knowledge, attitudes, and behaviors. Knowledge and attitude responses ranged from strongly disagree (1) to strongly agree (5) and behavior responses ranged from never (1) to always (5). Scores were summed across 3 questions within each subscale, so subscale scores ranged from 3-15 with 3 being the "worst" score and 15 being the "best" score. Population: For analysis of EHL questions, three subscales were created to assess knowledge, attitudes and behaviors related to EHL. Ordinal Likert scale responses were summed within the three subscales to create an approximately continuous variable for each. One participant had missing data for each of the knowledge and attitudes scales and 3 participants had missing data for the behaviors subscale.
  Scores on a Likert scale
    Knowledge subscale: number analyzed (Participants) | 433
    Knowledge subscale | 14.32 (0.85)
    Attitudes subscale: number analyzed (Participants) | 433
    Attitudes subscale | 13.03 (1.54)
    Behaviors subscale: number analyzed (Participants) | 431
    Behaviors subscale | 12.09 (2.03)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Endocrine Disrupting Chemical (EDC) Levels as Measured by the Post-intervention Value Minus the Baseline Value.
Description: Urine samples collected pre- and post-intervention to measure changes in EDC levels
Time Frame: Outcomes will be assessed at baseline (0-4 weeks) and up to 24 weeks for post-intervention
Population: 55 participants returned valid baseline and post-intervention urine samples for analysis. Values shown were adjusted for specific gravity. 7 participants had missing data for one or more variables necessary for the analysis (baseline, follow-up or specific gravity).
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Mobile EDC Reduction Program
Number analyzed (Participants) | 55
ng/ml
  methylparaben: number analyzed (Participants) | 48
  methylparaben | 5.83 (156.71)
  propylparaben | 18.43 (105.85)
  monobutyl phthalate | 56.94 (117.48)
  monoethyl phthalate | 75.30 (556.90)
  mono-(2-ethyl-5-carboxypentyl) phthalate | -3.47 (20.50)
Statistical Analysis 1: Comparison: Mobile EDC Reduction Program; Test type: Other; p < 0.05, t-test, 1 sided

2. Secondary Outcome: Changes in Environmental Health Literacy Using the Environmental Literacy Survey
Description: Validated survey on environmental health literacy will be conducted at baseline and upon completion of the second test. The surveys will be compared for changes. The EHL survey was adapted from the "General Environmental Health Scale" and was titled "Environmental Health Literacy Scale" with three subscales: knowledge, attitudes, and behaviors. Knowledge and attitude responses ranged from strongly disagree (1) to strongly agree (5) and behavior responses ranged from never (1) to always (5). Scores were summed across 3 questions within each subscale resulting in a range of 3 (worse) to 15 (better) for each subscale.
Time Frame: Outcomes will be assessed at baseline (0-4 weeks) and up to 24 weeks for post-intervention. Change scores are reported as the post-intervention subscale score minus the baseline score.
Population: For analysis of EHL questions, three subscales were created to assess knowledge, attitudes and behaviors related to EHL. Ordinal Likert scale responses were summed within the three subscales to create an approximately continuous variable for each, ranging from 3 (worse) to 15 (better). A positive change score reflecting higher post-intervention values is better. Two participants had missing data for the knowledge and attitude subscales and three had missing data for the behaviors subscale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile EDC Reduction Program
Number analyzed (Participants) | 174
units on a scale
  EHL Knowledge subscale: number analyzed (Participants) | 172
  EHL Knowledge subscale | -0.16 (1.13)
  EHL attitudes subscale: number analyzed (Participants) | 172
  EHL attitudes subscale | -0.14 (1.54)
  EHL behaviors subscale: number analyzed (Participants) | 171
  EHL behaviors subscale | 0.39 (1.70)
Statistical Analysis 1: Comparison: Mobile EDC Reduction Program; Paired samples t-tests were run to compare whether EHL knowledge, attitudes and behavior changed after the intervention. EHL scores were expected to increase between pre and post testing; Test type: Other; p < 0.05, paired samples t-test

ADVERSE EVENTS:
Time Frame: The intervention, from time of the first survey and urinalysis to the last, was typically 8 weeks.
Arm/Group | Mobile EDC Reduction Program
All-Cause Mortality (participants affected / at risk) | 0/434
Serious Adverse Events (participants affected / at risk) | 0/434
Other Adverse Events (participants affected / at risk) | 0/434

LIMITATIONS AND CAVEATS:
The lack of specificity and sensitivity in the EHL survey was a limitation of this study.

The difficulty in assessing low levels of EDC metabolites was also a challenge, as the current EDC testing panel has high detection limits for some of the metabolites.

The high attrition rate for the second urine test was also a problem, likely due to a long lag time without enough engagement and insufficient incentives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT05780047/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT05780047/SAP_001.pdf
  • Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT05780047/ICF_002.pdf